CLINICAL TRIAL: NCT02543944
Title: Improving Treatment Outcomes for Prescription Opioid Dependence
Acronym: GBN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 203970; R01DA039088 (NIH)
Record Dates: First submitted 2015-08-25; First posted 2015-09-07 (Estimated); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-05

CONDITIONS: Drug Dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Gabapentin; Buprenorphine; Clonidine; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin started on day 3 of week 1, increased up to a maximum dose of 800 mg BID by day 3 of week 2 and maintained for 2 weeks followed by 5-day taper.
  Buprenorphine (BUP) stabilization up to 12 mg (day 2 of week 1) then a 10-day BUP taper by the end of week 3.
  During week 4, detoxed subjects get 0.1 mg of clonidine followed by oral naltrexone (NTX) at 6.25 mg and another 6.25 mg (day 1), 25 mg (day 2) and 50 mg (day 3) then depot NTX injection (later on day 3 or day 4).
  Interventions: Drug: Gabapentin; Drug: Buprenorphine; Drug: Clonidine; Drug: Naltrexone (oral); Drug: Naltrexone (depot)
- Placebo (Placebo Comparator): Participants in this arm begin receiving placebo (microcrystalline cellulose) in twice daily capsules on day 3 of week 1 and continue to do so through the beginning of week 5.
  Buprenorphine (BUP) stabilization up to 12 mg (day 2 of week 1) then a 10-day BUP taper by the end of week 3.
  During week 4, detoxed subjects get 0.1 mg of clonidine followed by oral naltrexone (NTX) at 6.25 mg and another 6.25 mg (day 1), 25 mg (day 2) and 50 mg (day 3) then depot NTX injection (later on day 3 or day 4).
  Interventions: Drug: Buprenorphine; Drug: Clonidine; Drug: Naltrexone (oral); Drug: Naltrexone (depot); Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — N-type calcium channel blocker being examined for its potential efficacy to alleviate opioid withdrawal during buprenorphine-assisted detoxification and transition to depot naltrexone.
  Arms: Gabapentin
Drug: Buprenorphine — All participants are stabilized on buprenorphine and then undergo a 10 day taper off buprenorphine.
Drug: Clonidine — All participants who successfully taper off buprenorphine receive Clonidine (0.1 mg) prior to induction onto oral naltrexone.
Drug: Naltrexone (oral) — All participants receive increasing doses of oral naltrexone over a 3 day period (day 1: 6.25 and 6.25 mg; day 2: 25 mg; day 3: 50 mg)
Drug: Naltrexone (depot) — All participants who tolerate oral naltrexone at 50 mg will receive the naltrexone injection on either the same day as the 50 mg dose or the day after.
Drug: Placebo — Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Overall, this proposal seeks to improve treatment strategies for the significant public health problem of prescription opioid dependence by determining whether gabapentin, a non-narcotic pharmaceutical agent with minimal abuse potential and preliminary efficacy, will be effective in ameliorating withdrawal symptoms, craving and illicit drug use in prescription opioid dependent participants undergoing a 10-day detoxification from buprenorphine. In addition, the acceptability and feasibility of transitioning to depot naltrexone therapy will also be determined. If successful, this study would provide data to support further development of gabapentin as a pharmacological tool for improved outcomes during opioid detoxification as well as an integrated outpatient approach for treating prescription opioid dependence.

DETAILED DESCRIPTION:
Opioid dependence is a serious public health problem, particularly with the dramatic rise in prescription opioid abuse, but long-term opioid agonist maintenance with methadone or buprenorphine (BUP) may not be optimal for many prescription opioid abusers. Yet current opioid detoxification strategies are limited by high relapse rates and/or lack of efficacy in relieving subjective symptoms. In addition, antagonist maintenance with naltrexone (NTX), which may be an optimal longer-term strategy for this population, requires prior opioid detoxification and has been associated with relatively poor outcomes in heroin abusers. This application takes a novel, broad approach to address the problem of prescription opioid dependence by determining the 1) utility of adjunct gabapentin (GBP) during outpatient BUP detoxification to improve initial outcomes and 2) feasibility of transitioning prescription opioid -dependent patients to depot NTX following detoxification, which may improve longer-term outcomes. GBP, an N-type calcium channel blocker with low abuse potential, potentiates opioid analgesia, decreases both postoperative morphine consumption and movement-related pain, and reverses tolerance to the antinociceptive effects of morphine. GBP is also well tolerated and effective in reducing craving and illicit opioid use in pilot detoxification trials. The efficacy and tolerability of adjunct GBP during BUP-assisted detoxification and the feasibility of subsequent transition to depot NTX therapy in prescription opioid -dependent participants will be assessed. This 12-week, randomized, placebo-controlled clinical trial will determine the potential utility of adjunct GBP in 150 prescription opioid -dependent individuals undergoing outpatient BUP detoxification and whether transition to short-term depot NTX therapy is feasible. Our three specific aims are to determine (1) the efficacy and tolerability of GBP to reduce craving and illicit use of opioids in prescription opioid-dependent individuals undergoing outpatient BUP detoxification; (2) acceptability and feasibility of transition to, and short-term maintenance on, depot NTX following detoxification; and (3) prognosticators of completion of the BUP taper, successful induction onto depot NTX, symptomatology, and longer-term outcomes. Currently, the only Food and Drug Administration (FDA)-approved medications for the treatment of opioid withdrawal are the opioid agonists methadone and BUP, both of which have abuse liability, and NTX, which can produce low levels of withdrawal-like symptoms, especially early in treatment. Findings, if positive, will support further development of GBP as an adjunct medication as well as provide an integrated, seamless approach to outpatient prescription opioid-dependence treatment. Ultimately, this work could impact the addiction field by providing both procedural and pharmacological tools for treating prescription opioid dependence that significantly improve outpatient detoxification outcomes and markedly enhance access and transition to NTX therapy. This would shift clinical practice, establishing an effective adjunct regimen for BUP detoxification and an integrated approach for transition to NTX therapy. GBP may also be clinically useful for other situations where opioid withdrawal is a concern.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 18-65
2. be available to attend clinic 6 days a week for approximately 30-60 minutes per day during the first 4 3 weeks
3. fulfill Diagnostic Statistical Manual-5 criteria for moderate to severe opioid dependence. These criteria will be ascertained in the following manner: the physician will determine whether the individual is appropriate based on several clinical assessments that are routinely employed by methadone program physicians, including history and severity of opioid use, presence of track marks, prior treatment history, self-reported and/or observed signs and symptoms of opioid withdrawal. If any individual's degree of opioid dependence is questionable, that person will be excluded from further consideration as a participant.
4. submit a urine sample negative for benzodiazepines or barbiturates prior to starting the study.

Exclusion Criteria:

1. report having had a severe adverse reaction to study medications
2. have an unstable medical condition or stable medical condition that would interact with study medications or participation, including a current chronic pain or other medical condition that requires ongoing opioid agonist treatment (determined by physician assessment)
3. have a major psychiatric disorder (psychosis, schizophrenia, bipolar)
4. have major depression or anxiety disorder requiring psychoactive medication (as determined by physician)
5. physiological dependence on alcohol or drugs other than opioids, tobacco or marijuana (as determined by physician assessment)
6. are pregnant, plan to become pregnant or have inadequate birth control, if relevant
7. report ongoing use of over-the-counter or prescription drug (including Maalox) that would have major interaction with study drugs
8. have any of the following: liver function tests >3 times normal, blood urea nitrogen and Creatinine outside normal range; electrocardiogram abnormalities including but not limited to: bradycardia (<50 bpm); prolonged QT interval corrected for heart rate (>450 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block; pre-existing severe gastrointestinal narrowing (pathologic or iatrogenic).

Individuals with anxiety or depression will not be excluded unless they are taking prescription medication for their disorder under a physician's care or findings during screening indicate a need for immediate treatment determined by the study physician and/or the Columbia-Suicide Severity Rating Scale.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — University of Arkansas; Michael Mancino, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Ray A, Mancino MJ, Thostenson JD, Guise JB, Hendrickson HP, Nunes EV, Oliveto AH. Randomized, placebo-controlled trial of gabapentin during outpatient buprenorphine-assisted taper and transition to injectable naltrexone. Am J Drug Alcohol Abuse. 2025;51(6):761-775. doi: 10.1080/00952990.2025.2564757. Epub 2025 Dec 16. PMID 41401348

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Gabapentin started on day 3 of week 1, increased up to a maximum dose of 800 mg BID by day 3 of week 2 and maintained for 2 weeks followed by 5-day taper.
  Buprenorphine (BUP) stabilization up to 12 mg (day 2 of week 1) then a 10-day BUP taper by the end of week 3.
  During week 4, detoxed subjects get 0.1 mg of clonidine followed by oral naltrexone (NTX) at 6.25 mg and another 6.25 mg (day 1), 25 mg (day 2) and 50 mg (day 3) then depot NTX injection (later on day 3 or day 4).
  Gabapentin: N-type calcium channel blocker being examined for its potential efficacy to alleviate opioid withdrawal during buprenorphine-assisted detox and transition to depot naltrexone.
  Buprenorphine: All participants are stabilized on buprenorphine and then undergo a 10 day taper off buprenorphine.
  Clonidine: All participants who successfully taper off buprenorphine receive Clonidine (0.1 mg) prior to induction onto oral naltrexone.
  Naltrexone (oral): All participants receive increasing doses of oral naltrexone over a 3 day period (day 1: 6.25 and 6.25 mg; day 2: 25 mg; day 3: 50 mg)
  Naltrexone (depot): All participants who tolerate oral naltrexone at 50 mg will receive the naltrexone injection on either the same day as the 50 mg dose or the day after.
- Placebo: Participants in this arm begin receiving placebo (microcrystalline cellulose) in twice daily capsules on day 3 of week 1 and continue to do so through the beginning of week 5.
  Buprenorphine (BUP) stabilization up to 12 mg (day 2 of week 1) then a 10-day BUP taper by the end of week 3.
  During week 4, detoxed subjects get 0.1 mg of clonidine followed by oral naltrexone (NTX) at 6.25 mg and another 6.25 mg (day 1), 25 mg (day 2) and 50 mg (day 3) then depot NTX injection (later on day 3 or day 4).
  Buprenorphine: All participants are stabilized on buprenorphine and then undergo a 10 day taper off buprenorphine.
  Clonidine: All participants who successfully taper off buprenorphine receive Clonidine (0.1 mg) prior to induction onto oral naltrexone.
  Naltrexone (oral): All participants receive increasing doses of oral naltrexone over a 3 day period (day 1: 6.25 and 6.25 mg; day 2: 25 mg; day 3: 50 mg)
  Naltrexone (depot): All participants who tolerate oral naltrexone at 50 mg will receive the naltrexone injection on either the same day as the 50 mg dose or the day after.
  Placebo: Microcrystalline cellulose
Period: Phase 1: GBN/BUP Induction and BUP Detox
Arm/Group | Gabapentin | Placebo
Started | 60 | 57
Completed | 41 | 34
Not Completed | 19 | 23
Period: Phase 2: Transition From BUP to XR-NTX
Arm/Group | Gabapentin | Placebo
Started | 33 | 29
Completed | 12 | 12
Not Completed | 21 | 17
Period: Phase 3: XR-NTX Maintenance
Arm/Group | Gabapentin | Placebo
Started | 12 | 12
Completed | 7 | 3
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (8.3) | 32.5 (7.3) | 32.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 32 | 32 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 57 | 53 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 52 | 50 | 102
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 57 | 117
Education Level [Count of Participants; unit: Participants] — Level of education achieved on a categorical scale
  Participants
    Less than High School | 8 | 4 | 12
    High School/Some College/Vocational School | 43 | 46 | 89
    College Degree or higher | 8 | 5 | 13
    Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Detoxification Phase: Changes in Percent of Illicit Opioid-positive Urine Samples Over Time
Description: Thrice weekly urine samples obtained during weeks 1-3; data include assessments from week 1 day 1 through week 4 day 1 (up to 10 total samples per participant)
Time Frame: Week 1 day 1 (study entry) through Week 4 day 1 (first day of NTX transition)
Population: those starting on study medication
Measure: Mean (Standard Deviation); unit: percentage of urine positive samples
Units Other Than Participants: urine samples
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 60 | 57
Number analyzed (urine samples) | 455 | 421
percentage of urine positive samples | 35.0 (36.7) | 41.6 (38.5)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.77, Regression, Logistic; Risk Ratio (RR) = -0.0944, 95% CI 2-sided [-0.72 to 0.53], Standard Error of Mean 0.32

2. Secondary Outcome: NTX Transition Initiation
Description: % of Participants who completed the detox and started the NTX transition
Time Frame: 3 days (wk 4 day 1 - week 4 day 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 41 | 34
Participants | 33 | 29
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.58, Chi-squared; Odds Ratio (OR) = 0.3

3. Secondary Outcome: Vivitrol Injection Receivers
Description: % of participants starting the NTX transition who received Vivitrol injection
Time Frame: 5 days (week 4 day 1 to week 4 day 5)
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 33 | 29
Participants | 12 | 12
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.69, Chi-squared; Odds Ratio (OR) = 0.16

4. Secondary Outcome: Detox Phase Completers
Description: % of enrolled participants who completed the Detox Phase
Time Frame: 3 weeks (week 1-3)
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 60 | 57
Participants | 41 | 34
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.32, Chi-squared; Odds Ratio (OR) = .96

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/57
Other Adverse Events (participants affected / at risk) | 43/60 | 37/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=60) | Placebo (N=57)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain/soreness (Gastrointestinal disorders) | 2 (2) | 0 (0)
Loose, pale stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Urination changes (Renal and urinary disorders) | 6 (7) | 1 (1)
Bright colored urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Sedation/drowsiness (General disorders) | 8 (8) | 4 (4)
Listlessness/loss of energy (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3)
Weakness (General disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 2 (2)
Sleep disturbance/sleep walking (General disorders) | 1 (1) | 0 (0)
Restlessness (General disorders) | 1 (1) | 0 (0)
Muscle twitches/tremors (Nervous system disorders) | 5 (6) | 2 (2)
Tingling extremities (Nervous system disorders) | 1 (1) | 0 (0)
Muscle/skeletal pain/discomfort (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (2)
Tooth pain (General disorders) | 0 (0) | 1 (1)
Changes in equilibrium (General disorders) | 0 (0) | 2 (2)
Fall (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 7 (7) | 8 (8)
Dry mouth (General disorders) | 3 (3) | 2 (2)
Dry eyes (Eye disorders) | 0 (0) | 1 (1)
Burning sensation in eyes (Eye disorders) | 1 (1) | 0 (0)
Blood shot eye (Eye disorders) | 1 (1) | 0 (0)
Changes in vision (Eye disorders) | 3 (3) | 0 (0)
Changes in taste (General disorders) | 1 (1) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash on knees (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diagnosis of shingles (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bruising/laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hiccups (General disorders) | 1 (1) | 0 (0)
Elevated heart rate (Cardiac disorders) | 1 (1) | 2 (2)
Edema/swelling (General disorders) | 1 (1) | 1 (1)
Hot/cold sweats (General disorders) | 0 (0) | 1 (1)
Continuously hot all day (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Flu virus (Infections and infestations) | 1 (1) | 0 (0)
Sexual side effect (General disorders) | 1 (1) | 0 (0)
Auditory and visual hallucinations (General disorders) | 1 (1) | 0 (0)
Confusion/Disorientation (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 2 (2) | 1 (1)
Agitation (General disorders) | 1 (1) | 0 (0)
Anger (General disorders) | 1 (1) | 0 (0)
Symptoms of anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Symptoms of depression and/or anhedonia (Psychiatric disorders) | 1 (1) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Withdrawal symptoms (General disorders) | 13 (14) | 19 (25)
Withdrawal symptoms: not specified (General disorders) | 3 (3) | 1 (1)
Withdrawal sx: Related to dehydration (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Leg pain (General disorders) | 0 (0) | 2 (2)
Withdrawal sx: Muscle cramps (General disorders) | 1 (1) | 1 (1)
Withdrawal sx: Bone/muscle pain (General disorders) | 2 (2) | 2 (2)
Withdrawal sx: Stomach cramps (General disorders) | 2 (3) | 9 (9)
Withdrawal sx: Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6)
Withdrawal sx: Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Withdrawal sx: Diarrhea (Gastrointestinal disorders) | 2 (3) | 9 (9)
Withdrawal sx: Abdominal pain (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Loss of appetite (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0)
Withdrawal sx: Runny nose/sneezing and/or watery eyes (General disorders) | 1 (1) | 3 (3)
Withdrawal sx: Chills (General disorders) | 1 (1) | 1 (1)
Withdrawal sx: Hot/cold sweats (General disorders) | 0 (0) | 5 (6)
Withdrawal sx: Excessive sweating (General disorders) | 2 (2) | 3 (3)
Withdrawal sx: Fatigue (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Sedation (General disorders) | 0 (0) | 2 (2)
Withdrawal sx: Nodding off (General disorders) | 0 (0) | 0 (0)
Withdrawal sx: Insomnia (General disorders) | 2 (2) | 3 (3)
Withdrawal sx: Restlessness (General disorders) | 1 (1) | 3 (3)
Withdrawal sx: Yawning (General disorders) | 1 (1) | 2 (2)
Withdrawal sx: Stretching (General disorders) | 1 (1) | 0 (0)
Withdrawal sx: Muscle twiches/jerks (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Shakes/tremors (General disorders) | 2 (2) | 1 (1)
Withdrawal sx: Tingling extremities (General disorders) | 1 (1) | 0 (0)
Withdrawal sx: Headache (General disorders) | 1 (1) | 1 (1)
Withdrawal sx: Lightheaded (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Short of breath (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Dizziness (General disorders) | 1 (1) | 1 (1)
Withdrawal sx: Clammy feet/hands (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Gooseflesh (General disorders) | 0 (0) | 1 (1)
Withdrawal sx: Depression (General disorders) | 1 (1) | 1 (1)
Withdrawal sx: Anxiety (General disorders) | 1 (1) | 2 (2)
Withdrawal sx: Irritability (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT02543944/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT02543944/SAP_001.pdf
  • Informed Consent Form (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT02543944/ICF_002.pdf